CLINICAL TRIAL: NCT05557409
Title: ADVANCE-2: Addressing Dementia Via Agitation-Centered Evaluation 2: A Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of AXS-05 for the Treatment of Alzheimer's Disease Agitation
Brief Title: A Study to Assess the Efficacy and Safety of AXS-05 in Subjects With Alzheimer's Disease Agitation
Acronym: ADVANCE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXS-05-AD-304
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type; Alzheimer Disease; Agitation
Keywords: AD agitation; AXS-05; NMDA receptor antagonist; dextromethorphan; bupropion; Axsome; ADVANCE-2
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-05 (Experimental): Up to 5 weeks
  Interventions: Drug: AXS-05
- Placebo (Placebo Comparator): Up to 5 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-05 — AXS-05 tablets, taken twice daily
  Arms: AXS-05
Drug: Placebo — Placebo tablets, taken twice daily
  Arms: Placebo

SUMMARY:
This trial is a multi-center, double-blind, placebo-controlled, randomized study to evaluate the efficacy and safety of AXS-05 compared to placebo for the treatment of agitation associated with Alzheimer's disease.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 1:1 ratio for up to 5 weeks to be treated with AXS-05 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) based on the 2011 National Institute on Aging-Alzheimer Association (NIA-AA) criteria.
* Diagnosis of clinically significant agitation resulting from probable AD according to the International Psychogeriatric Association (IPA) provisional definition of agitation.

Exclusion Criteria:

* Patient has dementia predominantly of non-Alzheimer's type.
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 408 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | Up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (48):
- United States (46):
  - Clinical Research Site, Peoria, Arizona
  - Clinical Research Site, Tempe, Arizona
  - Clinical Research Site, Tucson, Arizona
  - Clinical Research Site, Canoga Park, California
  - Clinical Research Site, Long Beach, California
  - Clinical Research Site, Los Alamitos, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, West Covina, California
  - Clinical Research Site, Bonita Springs, Florida
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Greenacres City, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Kissimmee, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Gardens, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Pembroke Pines, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Augusta, Georgia
  - Clinical Research Site, College Park, Georgia
  - Clinical Research Site, Columbus, Georgia
  - Clinical Research Site, Wichita, Kansas
  - Clinical Research Site, Marrero, Louisiana
  - Clinical Research Site, Braintree, Massachusetts
  - Clinical Research Site, Flint, Michigan
  - Clinical Research Site, Rochester Hills, Michigan
  - Clinical Research Site, Troy, Michigan
  - Clinical Research Site, Chesterfield, Missouri
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, New Windsor, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Woodmere, New York
  - Clinical Research Site, Charlotte, North Carolina
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Cypress, Texas
  - Clinical Research Site, Mesquite, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Sugar Land, Texas
  - Clinical Research Site, Rutland, Vermont
  - Clinical Research Site, Arlington, Virginia
- Puerto Rico (2):
  - Clinical Research Site, Bayamón
  - Clinical Research Site, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://axsome.com/